CLINICAL TRIAL: NCT01950091
Title: Randomized Controlled Trial of Internet App to Self-Manage Occasional Low Back Pain
Brief Title: Internet App to Self-Manage Occasional Low Back Pain
Acronym: BackPain2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Center for Applied Science, Inc. (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, A. Blair Irvine, Research Scientist, Oregon Center for Applied Science, Inc.
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Back Pain II Study; R44AR054652 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-09-25 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Low Back Pain
Keywords: low back pain; internet; app; prevention; treatment
MeSH Terms: conditions — Low Back Pain; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FitBack on-line intervention (Experimental): On-line Fitback intervention: Self care for on-going pain; behaviors to lessen the chance of reoccurrence
  Interventions: Behavioral: FitBack on-line intervention
- Alternative website control (Active Comparator): Intervention is a Menu of links to 4 popular Websites offering back pain education
  Interventions: Other: Alternative Website Control
- Usual care control group (No Intervention): No contact; Control group

INTERVENTIONS:
Behavioral: FitBack on-line intervention — On-line Fitback intervention: Self care for on-going pain; behaviors to lessen the chance of reoccurrence
  Other Names: Fitback app
  Arms: FitBack on-line intervention
Other: Alternative Website Control — Intervention is a Menu of links to 4 popular Websites offering back pain education
  Arms: Alternative website control

SUMMARY:
Nonspecific low back pain (NLBP) is the diagnosis for 85% of low back pain sufferers with no underlying medical cause (e.g., herniated disc, spinal stenosis) that requires physician care. Treatment, however, is impractical for many physicians to implement during office visits, and there are relatively few providers for NLBP treatment that follow national pain control guidelines. This study evaluated the efficacy of an on-line intervention using desktop computers or mobile technology to help users self treat NLBP occurrences and to engage in activities to decrease future occurences.

DETAILED DESCRIPTION:
Methods. A total of 606 adults, 18 years of age and older were recruited, screened, and consented online. They were assessed on-line at baseline, at two months weeks, and at four months After the baseline assessments, participants were randomized into NLBP treatment (TX), alternative website control (AWC), and no-contact control groups. The TX and AWC groups received 8 weekly emails prompt to visit their respective experimental websites.

Add Details here.

ELIGIBILITY:
Inclusion Criteria:

* suffered low back pain in previous 3 months
* employed or family of employee

Exclusion Criteria:

* on-going medical care for low back pain
* positive response to questions about symptoms which medically disqualify potential participant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in responses to the Modified Oswestry Low Back Pain Disability Questionnaire | Baseline, 2 months, 4 months
  Back pain history: intensity, frequency, duration

SECONDARY OUTCOMES:
Change in responses to psycho-social measures (attitudes, knowledge, self efficacy, intentions); self treatment measures | baseline, 2 and 4 months
  Internally developed rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Blair Irvine, PhD, Principal Investigator — ORCAS Research Scientist

REFERENCES:
- [Derived] Irvine AB, Russell H, Manocchia M, Mino DE, Cox Glassen T, Morgan R, Gau JM, Birney AJ, Ary DV. Mobile-Web app to self-manage low back pain: randomized controlled trial. J Med Internet Res. 2015 Jan 2;17(1):e1. doi: 10.2196/jmir.3130. PMID 25565416